CLINICAL TRIAL: NCT04478474
Title: Cytomegalovirus (CMV) Viremia and Disease Occurrence in Pediatric Allogeneic Stem Cell Transplantation Recipients Following Ganciclovir Prophylaxis Until Day +100
Brief Title: Cytomegalovirus (CMV) Viremia and Disease Occurrence in Pediatric Allogeneic Stem Cell Transplantation Recipients
Status: Completed | Type: Observational
Sponsor: New York Medical College (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 14151
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Ganciclovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Eligible: Retrospective chart review of all pediatric patients who underwent allogeneic stem cell transplant between June 29, 2011 and December 31, 2019 at Westchester Medical Center (WMC). Children, adolescent, and young adult patients, ages 0-≤26 years, who have received an allogeneic stem cell transplantation on the pediatric bone marrow transplant service including matched unrelated donor, matched sibling donor, haploidentical donor, umbilical cord donor, who received ganciclovir prophylaxis for ≥14 days.
  Interventions: Drug: Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir — Type of allogeneic transplant, HLA match, graft manipulation, use of ATG and/or Campath, CMV status (donor and recipient), maximal acute GVHD stage and grade, CMV viremia/disease through day +100, days received ganciclovir prophylaxis, adverse events related directly or secondary to ganciclovir prophylaxis.
  Other Names: allogenic stem cell tranplatation

SUMMARY:
The primary objective is to determine the incidence of CMV viremia and disease in pediatric allogeneic stem cell transplantation recipients who received ganciclovir prophylaxis up until day +100 by retrospective analysis.

DETAILED DESCRIPTION:
This will be a single center, retrospective chart review of all pediatric patients who underwent allogeneic stem cell transplant between June 29, 2011 and December 31, 2019 at Westchester Medical Center (WMC). For this analysis, eligible patients will be identified through our transplantation database and clinical data collected through electronic medical record. This analysis will comprise of 100 pediatric allogeneic stem cell transplant recipients. CMV viremia will be defined as ≥2 CMV positive PCRs ≥500 copies and CMV disease will be defined as isolation of CMV in any body fluid or tissue specimen along with end-organ disease, as we have demonstrated.8 CMV viremia/disease will be evaluated through day +100 following allogeneic stem cell transplantation. Review of clinical records and collection of data with de-identified information will be performed. The study team will not access medical records (paper or electronic) directly. Medical records will be obtained through the Hospital's Health Information Management (HIM) department. HIM will query requested data / variables and provide a report / records of interest to Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective chart review of all pediatric patients who underwent allogeneic stem cell transplant between June 29, 2011 and December 31, 2019 at Westchester Medical Center (WMC).
* ages 0-≤26 years
* received an allogeneic stem cell transplantation on the pediatric bone marrow transplant service including matched unrelated donor, matched sibling donor, haploidentical donor, umbilical cord donor
* received ganciclovir prophylaxis for ≥14 days

Exclusion Criteria:

* None listed

Max Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescent, and young adult patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Ganciclovir | June 29, 2011 through December 31, 2019
  Ganciclovir will be safe, well tolerated, and effective to prevent CMV viremia and/or decrease in pediatric allogeneic stem cell transplant recipients.
CMV viremia and disease in pediatric allogenic SCT recipients | June 29, 2011 through December 31, 2019
  The primary objective is to determine the incidence of CMV viremia and disease in pediatric allogeneic stem cell transplantation recipients who received ganciclovir prophylaxis up until day +100 by retrospective analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Medical College, Valhalla, New York, United States

REFERENCES:
- [Background] Klejmont LM, Mo X, Milner J, Harrison L, Morris E, van de Ven C, Cairo MS. Risk Factors Associated with Survival Following Ganciclovir Prophylaxis through Day +100 in Cytomegalovirus At-Risk Pediatric Allogeneic Stem Cell Transplantation Recipients: Development of Cytomegalovirus Viremia Associated with Significantly Decreased 1-Year Survival. Transplant Cell Ther. 2024 Jan;30(1):103.e1-103.e8. doi: 10.1016/j.jtct.2023.09.025. Epub 2023 Oct 6. PMID 37806447